CLINICAL TRIAL: NCT03209466
Title: Standard Management and Chlorhexidine Gluconate Solution at 0.125% Versus Standard Management and Physiological Saline Sterile Solution for Healing Grade IIB Ulcers in Diabetic Foot Syndrome: Clinical Trial
Brief Title: Chlorhexidine Gluconate Solution at 0.125% vs Placebo for the Healing of Grade IIB Ulcers of Diabetic Foot
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Jose Antonio de Jesus Alvarez Canales, PhD, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHXDF
Record Dates: First submitted 2017-07-01; First posted 2017-07-06 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Diabetic Foot
Keywords: Chlorhexidine gluconate; Diabetic foot ulcer syndrome; Wound healing
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard management and Chlorhexidine gluconate at 0.125% (Experimental): Application every 24 hours, six weeks Intervention: Procedure: chlorhexidine gluconate
  Interventions: Drug: Chlorhexidine gluconate at 0.125%
- Standard management and physiological saline sterile solution (Placebo Comparator): Application every 24 hours, six weeks Intervention: Other: physiological saline sterile solution
  Interventions: Drug: Placebo Comparator with physiological saline sterile solution

INTERVENTIONS:
Drug: Chlorhexidine gluconate at 0.125% — Application every 24 hours, six weeks Intervention: Procedure: chlorhexidine gluconate
  Arms: Standard management and Chlorhexidine gluconate at 0.125%
Drug: Placebo Comparator with physiological saline sterile solution — Standard management and physiological saline sterile solution with application every 24 hours, six weeks Intervention.
  Arms: Standard management and physiological saline sterile solution

SUMMARY:
There is controversy regarding the utility of antiseptics in wound management for diabetic foot ulcer syndrome. The aim of this study is to assess chlorhexidine gluconate at 0.125% vs. saline solution to reduce the ulcerated area in patients with diabetic ulcer syndrome. A clinical trial model to evaluate modifications in size and area is proposed. Patients to be included will be those with diabetic foot ulcers Graded II accordingly to the University of Texas wound classification system.

DETAILED DESCRIPTION:
This study will be done in Hospital General de Leon

Population: People with diabetic foot syndrome grade IIb in Guanajuato Mexico

Universe: People with diabetes mellitus and diabetic foot syndrome in Guanajuato

Sample: Patients with diabetes mellitus over age of 18 years old, that present to the wound´s clinic of Hospital General Leon with diabetic foot ulcers classified as Texas IIB. This clinic provides services to patients in Guanajuato with diabetic foot syndrome, including them in a multidisciplinary management program.

Sample size calculation: A minimal sample of 35 patients for each arm of the study was calculated. Each study arm will be balanced considering the size. Potency was calculated at 0.8 and alpha value at 0-5, to detect a difference of 25% on the ulcer size.

Methodology:

Will be invited to participate in the study consecutive patients with diabetes mellitus presented with diabetic foot ulcers Graded II accordingly to the University of Texas wound classification system, in the area of Clinical wounds of Hospital General Leon between May and December 2017.

After explaining the study information and check it is understandable, the investigators provide the sheet to signed the informed consent.

Subsequently selected patients will be measure the ankle brachial index and determine the absence of vascular compromise.

Medical history with emphasis on analyzing clinical data, including the characteristics of the ulcer (type of exudate, measured surface area affected , type of tissue involved in the ulcer to its depth ) and biochemical parameters will be made.

Patients will be weighed and measured at the first visit and those who don't have biochemical data will be requested to collect this information in subsequent follow-up visits.

The participants will be then treated with the principles of the standard treatment, under the following criteria:

* Remove the ulcer exudate by spraying one of the two ingredients making mechanical drive for 5 minutes, or until completely negative to the visual evidence of exudate.
* Completely remove hyperkeratosis and devitalized tissue from the periphery of the ulcer with cutting material dissection with sterile dressing and drag, until visually eliminate the exudate.
* The treated area is dried.
* Two photographs at a distance of 20 cm perpendicular to the ulcer will be taken, covering a 1 square centimeter reference for measuring the area affected by diabetic foot ulcer syndrome.
* The solution will be applied in a blinded way to the ulcer and covered with sterile gauze for 24 hours.
* The patient will be instructed to continue treatment every 24 hours as follows:
* Sterile gauze will be removed and continuously irrigate for 5 seconds with the ingredient that was assigned.
* Undiscovered for 24 hours, until the next day irrigation gauze area will be placed. Also need to avoid contact with any surface over the affected area until the next assessment.
* Perform the same strategy for 24 hours, and on day 7 must go to the wound clinic to clinical evaluation.
* Every 7 days until complete 6 views, clinical evaluation is performed, irrigation with the selected ingredient and it will take 2 pictures at a distance of 20 cm perpendicular to the ulcer again, covering a reference of 1 square centimeter to measure the area affected by the diabetic foot ulcer syndrome.

Every week during the following 6 weeks, in the wound clinic consultation, it will be measured and gather information of the following elements:

* Ulcer area in square millimeters.
* Color of the ulcer.
* Type of exudate; turbid, serous.
* Type of tissue involved in the ulcer to its depth. If any patients have increased intensity of the signs and symptoms of diabetic foot syndrome, classified as a major step on the scale of ulcers Classification System of the University of Texas, perform analysis and comprehensive treatment will be redefined according to the suggestions of ulcer classification system of the University of Texas.

Cleaning material for the ulcer:

Ingredient 1: Preparation of spray application of chlorhexidine gluconate 0.125%.

Ingredient 2: Preparation of spray application of physiological saline sterile solution.

Method of application of ingredients as described previously. Method of randomization: will be effected since the fabrication of the ingredient by assigning a code number to each of the bottles that contained. Those bottles will have identical presentations, and will balance for the sample size. The code will not be known by the patient, observer and analyst. Only be known by one of the advisors.

Statistical methods:

The description of the data, in the case of non-numerical variables will be performed by reporting proportions and confidence interval of 95 % (95 %) in the case of numerical variables, the description will be made based on averages and standard deviation or medians and Q1- Q3 range, depending on the result of the Kolmogorov-Smirnov test to evaluate the Gaussian distribution of the data.

Comparison of numerical variables were not performed by Chi square test. Comparison of the rates of reduction in the size of ulcers of diabetic foot syndrome for both treatments will be based on the t test for independent samples or by Kruskal- Wallis test, depending on data distribution.

In all cases be considered as the significance level alpha value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients of both sex over age of 18 years old with diabetes mellitus that present an ulcer caused by diabetic foot syndrome with an extension from skin to tendon or join capsule and infected, classified as Texas IIB.

Exclusion Criteria:

* Patients lost to follow up and those that voluntary leave the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Ulcerated area | Up to 6 weeks
  area of diabetic foot ulcer measured with photographic register using a visual control of dimensions and a dedicated software for measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro E Macias, MD, Study Director — Universidad de Guanajuato
Locations (1):
- Universidad de Guanajuato, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No
None IPD will be share; only group data analyzed

REFERENCES:
- [Background] Frykberg RG, Zgonis T, Armstrong DG, Driver VR, Giurini JM, Kravitz SR, Landsman AS, Lavery LA, Moore JC, Schuberth JM, Wukich DK, Andersen C, Vanore JV; American College of Foot and Ankle Surgeons. Diabetic foot disorders. A clinical practice guideline (2006 revision). J Foot Ankle Surg. 2006 Sep-Oct;45(5 Suppl):S1-66. doi: 10.1016/S1067-2516(07)60001-5. PMID 17280936
- [Result] Boulton AJ, Vileikyte L, Ragnarson-Tennvall G, Apelqvist J. The global burden of diabetic foot disease. Lancet. 2005 Nov 12;366(9498):1719-24. doi: 10.1016/S0140-6736(05)67698-2. PMID 16291066
- [Result] Stewart PS, Costerton JW. Antibiotic resistance of bacteria in biofilms. Lancet. 2001 Jul 14;358(9276):135-8. doi: 10.1016/s0140-6736(01)05321-1. PMID 11463434